CLINICAL TRIAL: NCT00442663
Title: Randomized Trial of Transcervical Foley Catheter With and Without Extra-Amniotic Saline Infusion for Labor Induction
Brief Title: Trial of Foley Catheter With and Without Extra-Amniotic Saline Infusion for Labor Induction
Acronym: FOLEYEASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F050629003
Record Dates: First submitted 2007-02-28; First posted 2007-03-02 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Labor Induction; Cervical Ripening
Keywords: Labor Induction; Cervical Ripening; Foley Catheter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Transcervical Foley Catheter
Device: Transcervical Foley Catheter with an EASI

SUMMARY:
The purpose of this study is to compare the efficacy of a transcervical Foley catheter with and without extra-amniotic saline infusion (EASI) for priming the cervix for labor.

DETAILED DESCRIPTION:
In the United States, labor inductions have increased from 11% of all pregnancies in 1989 to 21% in 2004. Although the indications for labor induction vary, labor inductions as an obstetrical practice are associated with an increased risk of Cesarean delivery. As such, the rise in labor inductions has been paralleled by a rise in the cesarean rate to an all time high of 30%. The risk of cesarean can be mitigated with the use of cervical ripening agents in the setting of an unfavorable cervix. Both pharmacological ripening agents and mechanical methods are currently available for cervical priming. Methods available for mechanical dilation include, but are not limited to transcervical foley catheter alone and transcervical foley catheter with an extra-amniotic saline infusion or EASI. The potential advantage of EASI to transcervical foley catheter alone is the promotion of endogenous prostaglandin release by membrane stripping and supplying additional mechanical force. It may be disadvantageous by increasing the risk of chorioamnionitis or by diluting the prostaglandins that are released by membrane stripping. There have been two randomized trials comparing foley alone to foley with EASI. Because the results of these two trials are conflicting, we chose to conduct a randomized clinical trial of foley catheter compared to foley catheter with an EASI for labor induction and cervical ripening in women with an unfavorable cervix.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* 24-42 weeks of gestation
* Cephalic presentation
* Intact membranes
* Bishop score of less than or equal to 6

Exclusion Criteria:

* Contraindications to labor
* Dead or severely anomalous fetus
* Spontaneous labor.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 170
Dates: Start 2003-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Time from the start of labor induction to delivery

SECONDARY OUTCOMES:
Secondary maternal outcomes included cesarean delivery, chorioamnionitis and endometritis. Neonatal outcomes included birthweight, Apgar scores and cord blood gas analysis

CONTACTS AND LOCATIONS:
Overall Officials: Monique G Lin, MD, Principal Investigator — University of Alabama at Birmingham; George Lu, MD, Principal Investigator — Obstetrix Medical Group of Kansas City; Patrick S Ramsey, MD, MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (4):
- United States (4):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Truman Medical Center, Kansas City, Kansas
  - Saint Luke's Hospital, Kansas City, Kansas
  - Greenville Hospital System, University Medical Center, Greenville, South Carolina

REFERENCES:
- [Background] Guinn DA, Davies JK, Jones RO, Sullivan L, Wolf D. Labor induction in women with an unfavorable Bishop score: randomized controlled trial of intrauterine Foley catheter with concurrent oxytocin infusion versus Foley catheter with extra-amniotic saline infusion with concurrent oxytocin infusion. Am J Obstet Gynecol. 2004 Jul;191(1):225-9. doi: 10.1016/j.ajog.2003.12.039. PMID 15295370
- [Background] Karjane NW, Brock EL, Walsh SW. Induction of labor using a foley balloon, with and without extra-amniotic saline infusion. Obstet Gynecol. 2006 Feb;107(2 Pt 1):234-9. doi: 10.1097/01.AOG.0000198629.44186.c8. PMID 16449106
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Lin MG, Reid KJ, Treaster MR, Nuthalapaty FS, Ramsey PS, Lu GC. Transcervical Foley catheter with and without extraamniotic saline infusion for labor induction: a randomized controlled trial. Obstet Gynecol. 2007 Sep;110(3):558-65. doi: 10.1097/01.AOG.0000278077.30890.87. PMID 17766600